CLINICAL TRIAL: NCT06900309
Title: Effectiveness of a Home-based Telehealth Exercise Program Using the Physitrack App on Adherence and Performance in Handball Players: A Randomized Controlled Pilot Study
Brief Title: Effectiveness of a Home-based Telehealth Exercise Program on Adherence and Performance in Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEU-029
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Handball players performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific exercise program (Experimental): 8 weeks specific exercise program. Plyomteric exercises
  Interventions: Other: Specific exercise program
- Control (Active Comparator): 8 weeks general exercise program
  Interventions: Other: General exercise program

INTERVENTIONS:
Other: Specific exercise program — An 8-weeks specific exercise program based on lower limb plyomteric exercises
  Arms: Specific exercise program
Other: General exercise program — An 8-weeks of general exercise program focused on whole-body exercises
  Arms: Control

SUMMARY:
The objective of this clinical trial is to determine whether Physitrack®, a telerehabilitation platform, improves players' adherence to exercise programs. The secondary objectives are to assess whether its use enhances players' jumping ability (speed, height, flight time) and to evaluate the usability of the Physitrack® application from the players' perspective, considering aspects such as ease of use and user satisfaction.

The main questions this study aims to answer are:

Do exercise programs conducted through an online telemedicine platform achieve good adherence among handball players? Do exercise programs carried out via this telerehabilitation platform improve performance in vertical jumping? Do exercise programs performed using this platform provide good usability and user satisfaction results? To answer these questions, researchers will compare two groups following different exercise programs. The study will analyze whether, in addition to improving adherence, a specific program designed to enhance vertical jumping yields better results compared to a more general exercise program.

Participants:

Will perform a vertical jump test using force plates. Must follow the assigned eight-week exercise program according to randomization.

Will repeat the vertical jump test at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Men over 18 years old who are part of the Móstoles Handball Club team

Exclusion Criteria:

* Injured players at the start of the study and players who do not wish to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Percentage of adherence to the exercise program | From enrollment to the end of the program at 8 weeks
  Level of participation in the home exercise program through the Physitrack tele-rehabilitation platform measured as a percentage of program adherence

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Garcia-Catalan, Study Director — USP CEU University
Locations (1):
- USP CEU University, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: June 2025-June2028

REFERENCES:
- [Background] Balsalobre-Fernandez C, Varela-Olalla D. The Validity and Reliability of the My Jump Lab App for the Measurement of Vertical Jump Performance Using Artificial Intelligence. Sensors (Basel). 2024 Dec 10;24(24):7897. doi: 10.3390/s24247897. PMID 39771636
- [Background] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Background] Bennell KL, Lawford BJ, Metcalf B, Mackenzie D, Russell T, van den Berg M, Finnin K, Crowther S, Aiken J, Fleming J, Hinman RS. Physiotherapists and patients report positive experiences overall with telehealth during the COVID-19 pandemic: a mixed-methods study. J Physiother. 2021 Jul;67(3):201-209. doi: 10.1016/j.jphys.2021.06.009. Epub 2021 Jun 9. PMID 34147399
- [Background] Chang P, Engle J. Telemedicine and Virtual Interventions in Cancer Rehabilitation: Practical Application, Complications and Future Potentials. Curr Oncol Rep. 2024 Dec;26(12):1600-1605. doi: 10.1007/s11912-024-01612-8. Epub 2024 Nov 6. PMID 39503989
- [Background] Fristrup B, Krustrup P, Kristensen KH, Rasmussen S, Aagaard P. Test-retest reliability of lower limb muscle strength, jump and sprint performance tests in elite female team handball players. Eur J Appl Physiol. 2024 Sep;124(9):2577-2589. doi: 10.1007/s00421-024-05470-x. Epub 2024 Apr 9. PMID 38592403
- [Background] Satkunskiene D, Skarbalius A, Kniubaite A, Mickevicius M, Snieckus A, Rutkauskas S, Kamandulis S. Hamstring stiffness and injury risk factors during the handball season in female players. Appl Physiol Nutr Metab. 2024 Feb 1;49(2):190-198. doi: 10.1139/apnm-2023-0005. Epub 2023 Oct 11. PMID 37820386
- [Background] Badby AJ, Mundy PD, Comfort P, Lake JP, McMahon JJ. The Validity of Hawkin Dynamics Wireless Dual Force Plates for Measuring Countermovement Jump and Drop Jump Variables. Sensors (Basel). 2023 May 17;23(10):4820. doi: 10.3390/s23104820. PMID 37430733
- [Background] Dos'Santos T, Evans DT, Read DB. Validity of the Hawkin Dynamics Wireless Dual Force Platform System Against a Piezoelectric Laboratory Grade System for Vertical Countermovement Jump Variables. J Strength Cond Res. 2024 Jun 1;38(6):1144-1148. doi: 10.1519/JSC.0000000000004785. PMID 38781471
- [Background] Jaksic D, Maricic S, Maksimovic N, Bianco A, Sekulic D, Foretic N, Drid P. Effects of Additional Plyometric Training on the Jump Performance of Elite Male Handball Players: A Systematic Review. Int J Environ Res Public Health. 2023 Jan 30;20(3):2475. doi: 10.3390/ijerph20032475. PMID 36767841
- [Background] Anicic Z, Janicijevic D, Knezevic OM, Garcia-Ramos A, Petrovic MR, Cabarkapa D, Mirkov DM. Assessment of Countermovement Jump: What Should We Report? Life (Basel). 2023 Jan 9;13(1):190. doi: 10.3390/life13010190. PMID 36676138
- [Background] Manchado C, Tortosa Martinez J, Pueo B, Cortell Tormo JM, Vila H, Ferragut C, Sanchez Sanchez F, Busquier S, Amat S, Chirosa Rios LJ. High-Performance Handball Player's Time-Motion Analysis by Playing Positions. Int J Environ Res Public Health. 2020 Sep 17;17(18):6768. doi: 10.3390/ijerph17186768. PMID 32957441
- [Background] Suso-Marti L, La Touche R, Herranz-Gomez A, Angulo-Diaz-Parreno S, Paris-Alemany A, Cuenca-Martinez F. Effectiveness of Telerehabilitation in Physical Therapist Practice: An Umbrella and Mapping Review With Meta-Meta-Analysis. Phys Ther. 2021 May 4;101(5):pzab075. doi: 10.1093/ptj/pzab075. PMID 33611598